CLINICAL TRIAL: NCT00033436
Title: A Multicenter Randomized Trial of Radical Radiotherapy With Carbogen in the Radical Treatment of Locally Advanced Bladder Cancer
Brief Title: Radiation Therapy With or Without Carbogen and Niacinamide in Treating Patients With Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mount Vernon Cancer Centre at Mount Vernon Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000069283; MTVERNHOSP-BCON; EU-20051
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2002-12

CONDITIONS: Bladder Cancer
Keywords: stage I bladder cancer; stage II bladder cancer; stage III bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Niacinamide; carbogen; Radiotherapy

INTERVENTIONS:
Dietary Supplement: niacinamide
Drug: carbogen
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as carbogen and niacinamide may make tumor cells more sensitive to radiation therapy. It is not yet known whether radiation therapy is more effective with or without carbogen and niacinamide in treating patients who have bladder cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy with or without carbogen and niacinamide in treating patients who have locally advanced bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the 6-month cystoscopic response in patients with locally advanced transitional cell carcinoma of the bladder treated with radical radiotherapy with or without radiosensitization with carbogen and niacinamide.
* Compare the local failure-free and overall disease-specific survival of patients treated with these regimens.
* Compare the treatment-related morbidity, in particular acute and chronic bowel and bladder symptoms, in patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive radical radiotherapy once daily, 5 days a week, for 4-6.4 weeks. Patients also receive oral niacinamide once daily 1.5-2 hours before initiation of each radiotherapy dose and carbogen through a closed breathing system (face mask with a tight air seal or a mouthpiece with nasal clip) once daily beginning 5 minutes before initiation and continuing until completion of each radiotherapy dose.
* Arm II: Patients receive radiotherapy as in arm I. Quality of life is assessed at baseline; at 4 weeks; at 3, 6, and 12 months; and then annually for 4 years.

Patients are followed at 8 and 12 weeks; at 6, 9, and 12 months; and then every 6 months for 4 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 330 patients (165 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell carcinoma of the bladder

  * Muscle invasive carcinoma (stage T2 or T3) of any grade OR
  * High-grade (G3) superficial bladder carcinoma (T1) OR
  * Prostatic invasion (T4a)
* No squamous cell carcinoma or adenocarcinoma of the bladder
* No locally advanced T4b carcinoma
* No distant metastasis or enlarged pelvic lymph nodes on CT staging scan of the pelvis

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2 times normal

Renal:

* Creatinine no greater than 2 times normal

Cardiovascular:

* No ischemic heart disease or peripheral vascular disease requiring diuretics or angiotensin-converting enzyme inhibitors

Pulmonary:

* No concurrent respiratory disease with reduced respiratory drive that would preclude the delivery of 95% oxygen

Other:

* Capable of complying with a closed breathing system delivering carbogen through either a mask or a mouthpiece with nasal clip

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2000-10; Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Cystoscopic response at 6 months after initiation radiotherapy
Local failure-free survival
Overall disease-specific survival

SECONDARY OUTCOMES:
Treatment related morbidity (i.e., acute and chronic bowel and bladder symptoms)
Quality of life as assessed by FACT-BI scale at baseline, week 4, 3 months, 6 months, 12 months, and yearly thereafter for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Hoskin, MD, Study Chair — Mount Vernon Cancer Centre at Mount Vernon Hospital
Locations (14):
- United Kingdom (14):
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Derbyshire Royal Infirmary, Derby, England
  - Ipswich Hospital NHS Trust, Ipswich, England
  - Cookridge Hospital at Leeds Teaching Hospital NHS Trust, Leeds, England
  - Christie Hospital NHS Trust, Manchester, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Oldchurch Hospital, Romford, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales

REFERENCES:
- [Result] Hoskin PJ, Rojas AM, Saunders MI, Bentzen SM, Motohashi KJ; BCON investigators. Carbogen and nicotinamide in locally advanced bladder cancer: early results of a phase-III randomized trial. Radiother Oncol. 2009 Apr;91(1):120-5. doi: 10.1016/j.radonc.2008.10.001. Epub 2008 Nov 5. PMID 18992952
- [Derived] Choudhury A, Porta N, Hall E, Song YP, Owen R, MacKay R, West CML, Lewis R, Hussain SA, James ND, Huddart R, Hoskin P; BC2001 and BCON investigators. Hypofractionated radiotherapy in locally advanced bladder cancer: an individual patient data meta-analysis of the BC2001 and BCON trials. Lancet Oncol. 2021 Feb;22(2):246-255. doi: 10.1016/S1470-2045(20)30607-0. PMID 33539743